CLINICAL TRIAL: NCT05153954
Title: Quantitative ICG Fluorescence Angiography in Colorectal Surgery (QUANTICO): a Protocol for a Prospective, Standardized, Observational, Surgeon-blinded Multi-center Trial
Brief Title: Quantitative ICG Fluorescence Angiography in Colorectal Surgery
Acronym: QUANTICO
Status: Completed | Type: Observational
Sponsor: Zealand University Hospital (Other)
Collaborators: Perfusion Tech Aps (Unknown)
Responsible Party: Principal Investigator, Carolin Oppermann, Medical Doctor, PhD student, Zealand University Hospital
Other Study IDs: REG-046-2021
Record Dates: First submitted 2021-09-24; First posted 2021-12-10 (Actual); Last update posted 2024-12-03 (Actual); Status verified 2024-11

CONDITIONS: Colorectal Cancer; Anastomotic Leak
Keywords: indocyanine green; colon cancer; primary anastomosis; anastomotic perfusion; anastomotic leak
MeSH Terms: conditions — Colorectal Neoplasms; Anastomotic Leak; Colonic Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Colorectal cancer patients: Patients who can be treated with either PME or TME and receive a primary anastomosis during surgery.
  Interventions: Other: Quantitative Indocyanine Green Fluorescence Angiography

INTERVENTIONS:
Other: Quantitative Indocyanine Green Fluorescence Angiography — Quantitative analyse of ICG around the proximal/oral part of the anastomosis pre-formation of the primary anasomosis

SUMMARY:
Fluorescence angiography with indocyanine green (ICG-FA) has gained increased popularity in colorectal surgery to check perfusion to the newly-formed anastomotic area and decrease the rate of postoperative anastomotic leakage.

While qualitative ICG assessment has the advantage to be used instantly during the operative procedure, it does bear drawbacks (subjective assessment, dependent on factors like camera distance, ICG dose and white-light contamination).

The alternative is quantitative ICG assessment, which is performed by evaluating the time-intensity curve of the ICG-FA with an external analyzing software. The procedure is showing promising results, but the methodology is still reported very heterogeneously.

This study is a multi-center, prospective, standardized, surgeon-blinded observational trial. The key aspect of this study is the non-interventional design with blinding of both the qualitative and quantitative results from the ICG perfusion measurement, providing no chance of influencing the course of the operation. Assessment of perfusion will be performed postoperatively blinded to the outcome. Assessment of the pre-anastomotic area is intraoperatively performed by an image analysis software that then calculates a perfusion score based on an algorithm integrating relevant perfusion metrics. The primary outcome is the combined rate of early and late anastomotic complications within 90 days postoperatively.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years or older
* Capable of giving informed consent
* ASA Classification: status I-III
* Planned for PME or TME with minimally invasive approach and primary anastomosis
* Strong suspicion of or biopsy-verified sigmoid or rectal cancer Stage I-IV cancer

Exclusion Criteria:

* Known allergy to ICG or iodine
* Emergency procedure
* Pregnancy or if the patient is currently nursing
* Surgeons decide to do unblinded quantitative or qualitative ICG-FA

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study will include 115 participants undergoing elective resection with PME or TME for rectal or rectosigmoid cancer through a minimally invasive approach.
Sampling Method: Non-Probability Sample
Enrollment: 114 (Actual)
Dates: Start 2021-08-31 (Actual); Primary Completion 2024-08-31 (Actual); Study Completion 2024-11-28 (Actual)

PRIMARY OUTCOMES:
Postoperative anastomotic complications | 3 months
  combined rate of all anastomotic complications

SECONDARY OUTCOMES:
Number of participants with complications according to Clavien-Dindo Classification | 90 days
Number of participants with anastomotic leakage rate, severity (grade A-C) | 90 days
Number of participants with postoperative bleeding | 10 days
Number of participants with postoperative paralytic ileus | 90 days
  obstipation and intolerance of oral intake due to nonmechanical factors that disrupt the normal coordinated propulsive motor activity of the gastrointestinal tract following abdominal surgery
Number of participants with wound dehiscence | 1 month
  surgical complication in which a wound ruptures along a surgical incision
Comprehensive complications index | 90 days
Duration of surgery | 1 day
Reoperation rate | 1 month
Hospital readmission | 1 month
  Number of patients had have to be readmitted to the hospital due to postoperative complications
Length of hospital stay | 1 month
QT interval variability | 2 days
  Continuous ECG-monitoring intraoperatively and postoperatively

CONTACTS AND LOCATIONS:
Overall Officials: Ismail Gögenur, DMSc, MD, Principal Investigator — Department of Surgery, Zealand University Hospital; Niclas Dohrn, MD, Principal Investigator — Department of Surgery, Herlev Hospital; Mads Falk Klein, PhD, MD, Principal Investigator — Department of Surgery, Herlev Hospital
Locations (2):
- Denmark (2):
  - Department of Surgery, Zealand University Hospital, Køge, Region Sjælland
  - Department of Surgery, Herlev Hospital, Herlev

IPD SHARING:
Plan to Share IPD: No